CLINICAL TRIAL: NCT05899023
Title: Identifying Risk Factors for Poor Glycemic Control Among Emergency Department Patients and Improving Linkage to Outpatient Care
Brief Title: ED Diabetes Screening and Outpatient Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 23-00571
Record Dates: First submitted 2023-06-02; First posted 2023-06-12 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Diabetes Mellitus; Non Insulin Dependent Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telehealth Bridge Visits (Experimental): Patients in the experimental arm will receive post-emergency department telehealth bridge visits to connect ED patients with newly diagnosed diabetes to outpatient primary care.
  Interventions: Other: Telehealth Bridge Visits
- Control (Active Comparator): Patients in the control arm will receive standard of care.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Telehealth Bridge Visits — Patients will be scheduled for a telemedicine visit staffed by a family or internal medicine trained physician who will assess their understanding and answer any questions about the new diagnosis of diabetes, start initial conversations about how to improve their habits around diet and exercise, and discuss medication options for diabetes and, if appropriate, initiate treatment. At the end of the telemedicine visit, providers will attempt to address any difficulties that patients are experiencing in accessing primary care by providing an alternative contact for care or reaching out to a primary care doctor as necessary. If the patient experiences difficulties accessing a primary care provider based on their first telemedicine visit, then an additional telemedicine visit can be scheduled for the patient.
  Arms: Telehealth Bridge Visits
Other: Standard of Care — Standard of care currently includes calls from the site's follow-up center to see if patients received their HbA1c result, understood what their result meant, had any problems accessing medications prescribed or any difficulty scheduling an outpatient follow-up visit.
  Arms: Control

SUMMARY:
This goal of this NIH funded R01 study is to identify risk factors for not being able to follow-up for a new diagnosis of diabetes in the emergency department and improve linkage of these newly diagnosed patients to appropriate outpatient care. Its three aims will be accomplished through 1) a retrospective chart review of emergency department (ED) patients screened for diabetes, 2) a series of prospective qualitative interviews among ED patients with newly diagnosed diabetes who fail to follow-up for outpatient care, and 3) a simple randomized controlled trial to test the efficacy of telehealth bridge visits to connect ED patients with newly diagnosed diabetes to outpatient primary care.

ELIGIBILITY:
Inclusion Criteria:

* Emergency patient receiving lab tests with an initial HbA1c test result of ≥ 6.5%
* Residential address in New York City or Long Island
* Primary language is English or Spanish
* Able to provide informed consent

Exclusion Criteria:

* No prior history of diabetes
* No medical condition that would result in a spurious HbA1c test (e.g., sickle cell, recent blood loss)

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Percent of Patients who Complete at least One In-Person Follow-up Outpatient Visit | Up to Month 6 Post-Diagnosis
  A follow-up outpatient visit excludes the telehealth visits assigned to the experimental group. This outcome will be tracked using phone calls and data from Healthix, a regional health information exchange.

SECONDARY OUTCOMES:
Percent of Patients who Complete at least One Follow-Up Hemoglobin A1C (HbA1c) Test within 6 Months of Diagnosis | Up to Month 6 Post-Diagnosis
Percent of Patients who Complete at least One Follow-Up Hemoglobin A1C (HbA1c) Test within 12 Months of Diagnosis | Up to Month 12 Post-Diagnosis
Percent of Patients who Start on Diabetes Medications within 6 Months of Diagnosis | Up to Month 6 Post-Diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: David C. Lee, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared with researchers who provide a methodologically sound proposal upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: David.Lee@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: Researchers who provide a methodologically sound proposal will be granted access upon reasonable request. Requests should be directed to David.Lee@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.